CLINICAL TRIAL: NCT00074672
Title: Sensorimotor Gating Studies in Restless Legs Syndrome
Brief Title: Relationship Between Sensory and Motor Systems in Restless Leg Syndrome
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040059; 04-N-0059
Record Dates: First submitted 2003-12-17; First posted 2003-12-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-04-14

CONDITIONS: Restless Legs Syndrome
Keywords: Prepulse Inhibition; PPI; Dopamine; Sensorimotor Integration; Dopaminergic
MeSH Terms: conditions — Restless Legs Syndrome

SUMMARY:
This study will explore what occurs between sensory and motor systems in restless legs syndrome (RLS). Patients with RLS have uncomfortable sensations in the legs, usually in the evening or early part of the night. Most patients also have periodic involuntary leg movements. The condition tends to worsen over time, resulting in severe discomfort and sleep disturbances.

Healthy normal volunteers and patients with RLS between 18 and 80 years of age may be eligible for this study. All candidates will be screened with a medical history, physical and neurological evaluations, electroymogram (measure of muscle activity), overnight sleep study, electrocardiogram (ECG, measurement of the electrical activity of the heart), and blood and urine tests. They may also have brain or spine magnetic resonance imaging (MRI) or computerized tomography (CT) scans and a chest X-ray. Participants must stop taking all medications prohibited by the study for 2 days or more before the study starts and throughout its duration.

Participants will undergo prepulse inhibition tests to assess nervous system function. The participant sits comfortably in a quiet room. Several cables are attached to the face and legs using a special cream that conducts electrical signals through the cables to recording equipment. Nervous system activity is evaluated while the subject is at rest and after sensory stimulation (stimulating the nerves in the legs and face with a very brief electrical current of mild to moderate intensity). At times, the subject receives a short, mild sound stimulation delivered through earphones. The testing session takes 4 to 6 hours.

DETAILED DESCRIPTION:
Background - Restless leg syndrome (RLS), a condition affecting millions of Americans, is characterized by uncomfortable sensory symptoms relived by voluntary or involuntary movements. Objectives -To test our hypothesis that sensorimotor gating is deficient in RLS. Methods - In a controlled proof-of-principle clinical study, sensorimotor gating will be assessed through the use of validated electrophysiological tests of prepulse inhibition, in 17 adult patients with RLS and 17 matched healthy controls. Risks and benefits -Risks involved in this study are minimal, and deemed reasonable in relation to potential benefits. This investigation will lead to a better understanding of the pathophysiology of RLS.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects who meet all of the following inclusion criteria at screening will be eligible to participate in the study:

1. Male or female subjects aged 18 to 80.
2. For patients only, diagnosed with primary RLS based on the presence of a characteristic clinical history and the IRLSSG diagnostic criteria.
3. Normal physical and neurological examination.
4. Subject is willing to adhere to protocol requirements as evidenced by written, informed consent.
5. No clinically significant abnormalities on clinical chemistry or hematology examination at the pre-study medical evaluation.
6. Negative pre-study urine drug screen.

EXCLUSION CRITERIA:

Subjects meeting any of the following exclusion criteria will not be enrolled or will be immediately excluded from the study, as appropriate:

1. History of any medical condition that can reasonably be expected to compromise scientific integrity of the study;
2. Patient unwilling or unable to stop their usual mediations for RLS;
3. Subjects unable or unwilling to discontinue a prohibited concomitant medication
4. Subjects unwilling to sign an informed consent or to comply with protocol requirements.
5. Subjects with clinical and/or biological evidence of secondary RLS (e.g. renal failure (end-stage renal disease), iron deficient, anaemia or pregnancy at baseline).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2003-12-12; Study Completion 2009-04-14

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Walters AS. Toward a better definition of the restless legs syndrome. The International Restless Legs Syndrome Study Group. Mov Disord. 1995 Sep;10(5):634-42. doi: 10.1002/mds.870100517. PMID 8552117
- [Background] Silber MH. Restless legs syndrome. Mayo Clin Proc. 1997 Mar;72(3):261-4. doi: 10.4065/72.3.261. PMID 9070203
- [Background] Ondo W, Jankovic J. Restless legs syndrome: clinicoetiologic correlates. Neurology. 1996 Dec;47(6):1435-41. doi: 10.1212/wnl.47.6.1435. PMID 8960723